CLINICAL TRIAL: NCT04062331
Title: Clinical and Neurochemical Effects of Transcranial Magnetic Stimulation (TMS) in Multiple Sclerosis
Brief Title: Transcranial Magnetic Stimulation (TMS) in Multiple Sclerosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Isaac Tunez-Fiñana (Unknown); Eduardo Agüera-Morales (Unknown)
Responsible Party: Principal Investigator, Javier Caballero-Villarraso, Professor, Maimónides Biomedical Research Institute of Córdoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMTr-EMRR, ver - 3, 21/11/2017
Record Dates: First submitted 2019-08-01; First posted 2019-08-20 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
Keywords: clinical trial; multiple sclerosis; neurodegenerative diseases; transcranial magnetic stimulation; deep brain stimulation; neurochemistry
MeSH Terms: conditions — Multiple Sclerosis; Neurodegenerative Diseases | interventions — Transcranial Magnetic Stimulation; Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Phase I clinical trial, unicentric, controlled, randomised, single blind. Three arms.
  The patients included will be assigned under the 1:1:1 randomization formula, constituting three groups for the present study: 30 patients treated with natalizumab + white (placebo) + 30 patients treated with natalizumab + TMS (1 Hertz) + 30 patients treated with natalizumab + TMS (5 Hertz).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single-blind. Investigator who applies transcranial stimulation knows the kind of treatment (placebo, TMS 1 Hertz, TMS 5 Hertz). The patients don't know the frequency (measured Hertz) which TMS is running (0 Hertz= placebo, 1 Hertz, 5 Hertz) and the device and duration of sessions are the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo group (Placebo Comparator): This group will be under standard therapy (natalizumab) plus Transcranial Magnetic Stimulation (TMS) without any frequency (device doesn't running; it means, device turned off) but the same duration of sessions.
  Interventions: Drug: Placebos
- Group under TMS 1 Hertz treatment (Experimental): 1 Hertz group (1 Hertz ) will be under standard therapy (natalizumab) plus Transcranial Magnetic Stimulation (TMS) running with a frequency of 1 Hertz.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Group under TMS 5 Hertz treatment (Experimental): 5 Hertz group (5 Hertz ) will be under standard therapy (natalizumab) plus Transcranial Magnetic Stimulation (TMS) running with a frequency of 5 Hertz .
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — By means of the magnetic stimulator we induce a cerebral electric current that is able to obtain a motor potential in the first dorsal interosseous bone of the left hand.
  The intervention procedure consists of two steps: First step: Obtaining the Motor Evoked Threshold at Rest: Each patient, regardless of to the group to which they belong will have his/her threshold evoked motor calculated at rest, by stimulation of the right motor cortex, evoking electromyographic responses in the contralateral muscles. Second step: Administration of TMS: To calculate the motive threshold as the percentage of the same to which the treatment will have to be applied, a device equipped with a coil. The treatment will be administered for 5 consecutive days, with 3 weeks of rest, between each stimulation. To complete a treatment period of 14 months. The stimulation with TMS will be carried out every day in the same time slot for 5 consecutive days every 4 weeks, during a period of 14 months.
  Other Names: Deep Brain Stimulation; Deep Transcranial Magnetic Stimulation
  Arms: Group under TMS 1 Hertz treatment; Group under TMS 5 Hertz treatment
Drug: Placebos — Administration of Transcranial Magnetic Stimulation at 0 Hz (the patient will be only under drug standar therapy)
  Other Names: Sham group
  Arms: Placebo group

SUMMARY:
Background: Transcranial Magnetic Stimulation (TMS) is a technique based on the principles of electromagnetic induction. It applies pulses of magnetic radiation that penetrate the brain tissue, and it is a non-invasive, painless and practically innocuous procedure. Previous studies advocate the therapeutic capacity of TMS in several neurodegenerative and psychiatric processes, both in animal models and in human studies. Its uses in Parkinson's disease, Alzheimer's disease and in Huntington's chorea have shown improvement in the symptomatology and in the molecular profile, and even in the cellular density of the brain. Consequently, the extrapolation of these TMS results in the aforementioned neurodegenerative disease to other entities with etiopathogenic and clinical analogy would raise the relevance and feasibility of its use in multiple sclerosis (MS). The overall objective will be to demonstrate the effectiveness of the TMS in terms of safety and clinical improvement, as well as to observe the molecular changes in relation to the treatment.

Methods and design: Phase I clinical trial, unicentric, controlled, randomised, single blind. A total of 90 patients diagnosed with relapsing-remitting multiple sclerosis (RRMS) who meet all the inclusion criteria and do not present any of the exclusion criteria that are established and from which clinically evaluable results can be obtained. The patients included will be assigned under the 1:1:1 randomization formula, constituting three groups for the present study: 30 patients treated with natalizumab + white (placebo) + 30 patients treated with natalizumab + TMS (1 Hertz) + 30 patients treated with natalizumab + TMS (5 Hertz).

Discussion: Results of this study will inform on the efficiency of the TMS for the treatment of MS. The expected results are that TMS is a useful therapeutic resource to improve clinical status (main parameters) and neurochemical profile (surrogate parameters); both types of parameters will be checked.

DETAILED DESCRIPTION:
It is based on the hypothesis that the application of transcranial magnetic stimulation (TMS) at 1 Hertz or 5 Hertz in patients with relapsing-remitting multiple sclerosis (RRMS) implies a neuroprotective effect against the progression of the disease, resulting in a clinical improvement (attenuation of symptoms and signs, as direct measures of the therapeutic effect) and a biochemistry improvement (decrease of serum oxidative stress molecules and acute phase reactants, as indirect measures).

Along with the traditional techniques for measuring biochemical magnitudes, proteomic techniques would allow the identification (and subsequent validation) of molecules that are clearly different in situations of stability-relapse, presence-absence of therapeutic response, better-worse evolution. These molecules (in isolation or considering their characteristics together) could be useful as therapeutic targets or as useful biomarkers for diagnostic or prognostic use.

The main goal is to demonstrate the therapeutic effect of TMS in patients with MS by means of measurement of clinical changes according to the Expanded Disability Status Scale (EDSS). Consequently, the specific objectives are:

* To determine the consequences of the administration of TMS (1 Hertz/5 Hertz) in patients with MS, paying special attention to its clinical impact according to the MSFC scale (Multiple Sclerosis Functional Composite).
* To assess the effect of the application of TMS (1 Hertz/5 Hertz) on fatigue in people with MS, according to the FIS scale (Fatigue Impact Scale).
* To observe the effect of the application of TMS (1 Hertz/5 Hertz) on the degree of depression, according to the Beck scale.
* To study the impact of TMS (Hertz/5 Hz) on cognitive changes in patients with MS, in relation to the BRB scale (Brief Repeatable Battery of Neuropsychological Test).
* To identify the changes induced by the application of TMS (1 Hertz/5 Hertz) on neurochemical biomarkers, oxidative damage, acute phase reactants and in differential expression proteomic profiles, in patients affected by MS.
* To establish the possible associations between the parameters studied and the likely changes that may be observed in them after TMS therapy.

DESIGN:

Phase II clinical trial, unicentric, controlled, randomised, single blind. The patients included will be assigned under the 1:1:1 randomization formula, constituting three groups for the present study: 30 patients treated with natalizumab + white (placebo) + 30 patients treated with natalizumab + TMS (1 Hertz) + 30 patients treated with natalizumab + TMS (5 Hertz).

SELECTION OF SUBJECTS:

PATIENT SAMPLE TO STUDY.- 90 patients diagnosed with RRMS, who meet all the inclusion criteria and do not present any of the exclusion criteria that are established below and from which clinically evaluable results can be obtained.

VARIABLES TO STUDY:

Patients will be evaluated by:

1. Clinical activity of the disease: Expanded Disability Status Scale (EDSS).
2. Comprehensive clinical assessment of the disease: Multiple Sclerosis Functional Composite (MSFC).
3. Cognitive function: Brief Repeatable Battery of Neuropsychological Test (BRB).
4. Assessment of fatigue: Fatigue Impact Scale (FIS).
5. Depression assessment: Beck depression scale.
6. Radiological: Nuclear Magnetic Resonance (NMR) with and without contrast.
7. Complete blood count(with formula and count of red, white and platelet series) and Biochemistry (glucose, lipid profile, total proteins, albumin, transaminases, CK and LDH).
8. Biomarkers of oxidative damage: lipoperoxidation products and plasma carbonylated proteins.
9. Redox state of glutathione (glutathione (GSH), glutathione disulfide (GSSG) and GSH/GSSG ratio).
10. Levels of neurotrophic factors (BDNF and NGF).
11. Cytokines: TNFalpha.
12. Studies of proteomics with "equalisation" and further bioinformatic analysis.

POPULATIONS AND JUSTIFICATION OF THE CHOICE OF NATALIZUMAB AS A BASAL MEDICATION:

The feasibility analysis will be done by intention to treat, and will include all patients for whom investigators have some feasibility data.

Patients in the three RRMS groups are treated with natalizumab. It could have been decided to recruit those treated with another pharmacological therapy (such as alemtuzumab, being a more modern monoclonal antibody); however, natalizumab offers us four advantages:

i) Its idiosyncrasy of administration (intravenous) leads to the patient going to the hospital and undergoing a blood analysis, which facilitates obtaining the sample needed in the present study.

ii) It is the drug with which a greater number of patients with RRMS is currently being treated in our hospital, which makes it possible to maximise the possibilities of recruitment.

iii) Regarding the previous point, considering patients under the same treatment (pharmacological) allows us to homogenise the characteristics of the three groups of the sample recruited, which increases the internal and external validity of results.

iv) To the above the investigators can add that natalizumab is the drug with which the research group has the most experience.

POSSIBLE LOSS OF PATIENTS: RETIREMENT CRITERIA AND ANALYSIS OF ANTICIPATED WITHDRAWALS AND ABANDONMENTS:

A withdrawal is defined as the situation in which a subject included in the Clinical Trial ends his/her participation in it before completing the protocol in its entirety, independently of the circumstances that motivate the termination. Patients will interrupt their participation and will be removed from the clinical trial in any of these situations:

i) Presence of a serious adverse event since the patient's recruitment. ii) Clinical conditions of the patient that prevent his/her continuity. iii) Other reasons: protocol violation, lack of cooperation, revocation of informed consent, loss of follow-up.

The date and reason why a subject interrupts his/her participation in the Clinical Trial must be recorded in the Data Collection Notebook. The circumstance of the interruption should be notified immediately to the monitor and if this has been a Serious Adverse Event.

The patient has the full right to leave the study at any time and any patient can be removed from the study for any reason beneficial to his/her well-being. According to the standards of Good Clinical Practice (GCP), all patients who leave the study before the foreseen time will be recommended the best alternative treatment.

CONTINGENCY PLAN:

This has been planned from a preventive point of view. Therefore, before starting it was assumed up to 20% loss of patients' follow-up in the calculation of the sample size.

ETHICAL, SOCIAL, LEGAL AND ENVIRONMENTAL PROJECT IMPLICATIONS:

The proposed clinical trial will be conducted in accordance with the protocol following the standard procedures established at the participating hospital. Said trial will be carried out according to the recommendations for Clinical Trials and product evaluation in human research phase, which appear in the Declaration of Helsinki, reviewed in the successive world assemblies (WMA, 2008), and the current Spanish Legislation in the field of Clinical Trials (RD 1090/2015). The International Conference on Harmonization (ICH-GCP) standards (CPMP/ICH/135/95) will be followed. The Clinical Research Ethics Committee (CEIC) of Córdoba has already reviewed and approved the protocol and informed consent in December 2017, as well as the completion of the present clinical trial itself. Before carrying out any of the procedures specified in the protocol, the participating subject must sign and date the informed consent document approved by the CEIC.

In order to guarantee the confidentiality of the trial data, the original data will be kept in the hospital and will only be accessed by the researcher and his/her team of collaborators, the trial monitor and the CEIC of Córdoba, which is the body that would protect the present essay. The researcher will allow the audits and inspections of the Spanish or European Health Authorities.

The content of the data collection notebooks and the confidentiality of the data of each patient will be respected at all times. Appropriate procedures will be followed to ensure compliance with the provisions of Organic Law 15/99 of December 13 on the Protection of Personal Data. The documents generated during the study, will be protected from uses not allowed by people outside the investigation and, therefore, will be considered strictly confidential and will not be disclosed to other people.

Note 1: DESCRIPTION OF THE TREATMENT:

By means of the magnetic stimulator with the coil located in the primary motor cortex the investigators induce a cerebral electric current that is able to obtain a motor potential in the first dorsal interosseous bone (PID) of the left hand. The investigators will measure muscle stimulation by placing conventional surface electrodes connected to a device of evoked potentials. It is a Compound Muscle Action Potential (PAMC) that represents the sum of the action potentials of all the individual muscle fibres underlying the electrodes. For this, the electromyograph is programmed with the following parameters: A) Sensitivity: 50 uV; B) Frequency filter: between 2000 Khz and 1 Hz; C) Scan speed 10 ms / div; D) Digitised preamplification signs, and v) Surface electrodes are placed: active in the eminence of the dorsal interosseous muscle and reference in the dorsal bony prominence of the second finger.

The procedure will depend on the group to which the patient has been assigned. In groups 2 and 3, the investigators will place the probe from 8 to 3 centimetres in front of the vertex (Cz) medially and perpendicular to the craniocaudal axis.

Note 2: DETAILS OF THE PROCEDURE:

The intervention procedure consists of two steps:

First step: OBTAINING THE MOTOR EVOKED THRESHOLD AT REST: Each patient, regardless of to the group to which they belong will have his/her threshold evoked motor calculated at rest, by stimulation of the right motor cortex, evoking electromyographic responses (EMG) in the contralateral muscles, called motor evoked potentials (PEM).

Second step: ADMINISTRATION OF THE TRANSCRANIAL MAGNETIC STIMULATION: To calculate the motive threshold as the percentage of the same to which the treatment will have to be applied, a 'Rapid2 Magstim' device (Magstim Co.®, Whitland, Carmathenshire, Wales) equipped with a coil in eight of 70 mm, will be used. The selection of the specific point of stimulation in the somato-sensory area (SMA) will be sufficiently anterior to prevent the propagation of the impulse from triggering the muscular contraction of the shoulders, trunk and lower limbs. The treatment will be administered for 5 consecutive days, with 3 weeks of rest, between each stimulation. To complete a treatment period of 14 months (based on previous studies of the group in RRMS patients treated with natalizumab). In the case of the placebo group (patients with RRMS treated with natalizumab and placebo coil) patients will be stimulated with an inactive probe, the perception being indistinguishable.

The stimulation with TMS (or administration of placebo) will be carried out every day in the same time slot for 5 consecutive days every 4 weeks, during a period of 14 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with RRMS in their inflammatory forms who have completed a 14-dose treatment with natalizumab.
2. Normal analytical parameters, defined by: Leukocytes> 3000 / mcl, Neutrophils> 1500 / mcl, Platelets> 100000 / mcl, AST/ALT <2.5 IU / L, Creatinine <2.5 mg / dl.
3. Patients of both sexes aged between 18 and 60 years.
4. EDSS: between 3.0 and 6.5 points.
5. Patients who give their informed consent for participation in the clinical trial.
6. Women of childbearing potential must obtain negative results in a pregnancy test performed at the time of inclusion in the study and commit to using a medically approved method of contraception for the duration of the study.

Exclusion Criteria:

1. Any active or chronic infection, including HIV infection, or hepatitis B or C.
2. History of neoplasia (basal cell carcinoma of the skin and in situ carcinoma in remission are excluded for more than one year).
3. Life expectancy severely limited by other co-morbidities.
4. Endocrine disease such as diabetes, hyper or hypothyroidism.
5. Chronic inflammatory or autoimmune disease such as ulcerative colitis, Crohn's disease, systemic lupus erythematosus and any other form of connective tissue disease or chronic arthropathy.
6. Chronic obstructive pulmonary disease.
7. Severe psychiatric illnesses.
8. Hepatic, or renal, or cardiac dysfunction (including coronary heart disease and heart failure).
9. Chronic anaemia.
10. Pregnancy or risk of pregnancy (including refusal to use contraception).
11. Women in breastfeeding period.
12. Inability to undergo MRI scans.
13. Inability to grant written informed consent.
14. Taking lipid-lowering drugs and vitamin supplements.
15. Treatment with steroids and/or non-steroidal anti-inflammatories, or alcohol intake 40 hours before the blood extraction and/or development of the different tests.
16. Chronic alcoholism and/or abuse of drugs of abuse (sporadic or chronic).
17. Metallic implants in the head.
18. Cardiac pacemaker device.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical activity of the disease | up 1 year
  Expanded Disability Status Scale. Score from 0 (total absence of disability) to 10 (death due to multiple sclerosis).
Comprehensive clinical assessment of the disease | up 1 year
  Multiple Sclerosis Functional Composite. It consists of three tests: Timed 25-Foot Walk, 9-Hole Peg Test and Paced Auditory Serial Addition Task. Score measured as a function of time. The higher, the worse the patient's condition.
Cognitive function | up 1 year
  Brief Repeatable Battery of Neuropsychological Test. It consists of the selective reminding test, the 10/36 spatial recall test, the symbol digit modalities test, the paced auditory serial addition test and the word list generation test. A higher score means a better status in a person.

SECONDARY OUTCOMES:
Assessment of fatigue | up 1 year
  Fatigue Impact Scale. It is based on items derived from interviews with MS patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. It consists of 21 items. A higher score means a worse status in a person.
Depression assessment | up 1 year
  Beck depression scale It is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Score from 0 to 63 (0 is no depression and 30-63 interval means several depression).
Image analysis | through study completion, an average of 1 year
  Nuclear Magnetic Resonance with and without contrast
Lipoperoxidation molecules | through study completion, an average of 1 year
  malondialdehyde (ng/mL) and 4-hydroxynonenal (ng/mL)
Carbonylated proteins | through study completion, an average of 1 year
  carbonyl reductase (nmol/mL) and carbonyl (nmol/mL)
Complete blood count | through study completion, an average of 1 year
  Complete blood count (with formula and count of red, white and platelet series)
glucose | through study completion, an average of 1 year
  glucose (mg/dL)
Routine serum lipids | through study completion, an average of 1 year
  cholesterol (mg/dL) and triglycerides (mg/dL)
Routine serum proteins | through study completion, an average of 1 year
  total proteins (g/L) and albumin (g/L)
Transaminases | through study completion, an average of 1 year
  aspartate aminotransferase (AST) (IU/L) and alanine aminotransferase (AST) (IU/L)
creatine kinase (CK) | through study completion, an average of 1 year
  CK (mg/mL)
lactate dehydrogenase | through study completion, an average of 1 year
  LDH (mg/mL)

IPD SHARING:
Plan to Share IPD: Yes
To publish the protocol study and its results in Scientific Journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The protocol study may be published in the last quarter of 2019. The results could be published at the end of the study (about 2022).
Access Criteria: Throug the website of research group https://www.imibic.org/grupo/35 or after request it (by previous e-mail from one of investigators)

REFERENCES:
- [Derived] Aguera E, Caballero-Villarraso J, Feijoo M, Escribano BM, Conde C, Bahamonde MC, Giraldo AI, Paz-Rojas E, Tunez I. Clinical and Neurochemical Effects of Transcranial Magnetic Stimulation (TMS) in Multiple Sclerosis: A Study Protocol for a Randomized Clinical Trial. Front Neurol. 2020 Aug 11;11:750. doi: 10.3389/fneur.2020.00750. eCollection 2020. PMID 32849212